CLINICAL TRIAL: NCT03918408
Title: Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Collagen Cross-Linking in Eyes With Corneal Thinning Conditions
Brief Title: Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Cross-Linking
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pacific Clear Vision Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1005312
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Keratoconus, Unstable; Bacterial Keratitis; Ectasia of Cornea
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: Treatment of patients with disease
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized at outset
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulsed, accelerated (Experimental): 18 mW, 5 sec, 5 sec off, 10 minutes of illumination
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke ribofflavin solution
- Conventional (Active Comparator): 9 mW, continuous 10 minutes of illumination
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke ribofflavin solution

INTERVENTIONS:
Combination Product: PXL-330 Platinum device for crosslinking with Peschke ribofflavin solution — Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea
  Other Names: Corneal crosslinking

SUMMARY:
To determine whether the Peschke PXL-330 system is safe and effective in the treatment of corneal thinning conditions.

DETAILED DESCRIPTION:
Patients with progressive keratoconus, pellucid marginal degeneration, infectious keratitis, or at risk for post-refractive corneal ectasia will be recruited and undergo epithelial-on corneal crosslinking with the Peschke PXL-330 system using pulsed, accelerated energy delivery. Patients will undergo monitoring for 1 year, with serial measurements of corneal topography, visual acuity, intraocular pressure, and visual function questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Subjects who have one or both eyes that meet criteria 1 & 2 and 1 or more of the following criteria will be considered candidates for this study.

* 12 years of age or older
* Evidence of progressive keratoconus (based on the discretion of the physician as evidenced by an increase in astigmatism, asymmetry, or worsening vision in the last 3 or more months)
* Presence of central or inferior steepening.
* Axial topography consistent with keratoconus
* Presence of one or more findings associated with keratoconus such as:
* Fleischer ring
* Vogt's striae
* Decentered corneal apex
* Munson's sign
* Rizzutti's sign
* Apical Corneal scarring consistent with Bowman's breaks
* Scissoring of the retinoscopic reflex
* Crab-claw appearance on topography
* Steepest keratometry (Kmax) value ≥ 47.20 D
* I-S keratometry difference > 1.5 D on the Pentacam/Galilei/Orbscan/Cassini map or topography map
* Posterior corneal elevation >16 microns
* Thinnest corneal point <485 microns
* AvaGen (Avellino Labs) genetic testing keratoconus risk score of 67 or higher (high risk).
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits
* For Contact Lens Wearers Only: Removal of contact lenses for the required period of time prior to the screening refraction:
* Contact Lens Type Minimum Discontinuation Time:
* Soft: 1 Week
* Soft Extended Wear: 2 Weeks
* Soft Toric: 3 Weeks
* Rigid gas permeable: 2 Weeks per decade of wear
* Scleral Lenses
* Investigator Discretion [Discontinuation of scleral lenses not required unless there is clinical evidence of corneal hypoxia (e.g. corneal neovascularization) at time of screening]
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria (any of the following are reasons for exclusion):

* Eyes classified as either normal or atypical normal on the severity grading scheme.
* Corneal pachymetry at the screening exam that is <330 microns at the thinnest point in the eye(s) to be treated.
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:
* History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthomeoeba, etc.)
* Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure.
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
* Patients with active medical implants (e.g. cardiac pacemakers)'
* Patients who are aphakic/ pseudophakic

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Mean keratometry in diopters | 12 months
  Average keratometry across the anterior topography of the cornea computed by a validated Scheimpflug topographer

SECONDARY OUTCOMES:
Best corrected visual acuity | 12 months
  Measurement of best corrected visual acuity on the validated early-treatment diabetic retinopathy study scale

CONTACTS AND LOCATIONS:
Overall Officials: BALAMURALI AMBATI, MD, PhD, Principal Investigator — PCVI
Locations (1):
- Pacific Clear Vision Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be stored in a secure location. While summary outcomes data will be provided on request to other researchers and periodically at scientific conferences, protected health information will not.

REFERENCES:
- [Background] Caporossi A, Baiocchi S, Mazzotta C, Traversi C, Caporossi T. Parasurgical therapy for keratoconus by riboflavin-ultraviolet type A rays induced cross-linking of corneal collagen: preliminary refractive results in an Italian study. J Cataract Refract Surg. 2006 May;32(5):837-45. doi: 10.1016/j.jcrs.2006.01.091. PMID 16765803
- [Background] Caporossi A, Mazzotta C, Baiocchi S, Caporossi T. Long-term results of riboflavin ultraviolet a corneal collagen cross-linking for keratoconus in Italy: the Siena eye cross study. Am J Ophthalmol. 2010 Apr;149(4):585-93. doi: 10.1016/j.ajo.2009.10.021. Epub 2010 Feb 6. PMID 20138607
- [Background] Chatzis N, Hafezi F. Progression of keratoconus and efficacy of pediatric [corrected] corneal collagen cross-linking in children and adolescents. J Refract Surg. 2012 Nov;28(11):753-8. doi: 10.3928/1081597X-20121011-01. PMID 23347367
- [Background] Mazzotta C, Traversi C, Caragiuli S, Rechichi M. Pulsed vs continuous light accelerated corneal collagen crosslinking: in vivo qualitative investigation by confocal microscopy and corneal OCT. Eye (Lond). 2014 Oct;28(10):1179-83. doi: 10.1038/eye.2014.163. Epub 2014 Jul 25. PMID 25060847

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03918408/Prot_SAP_000.pdf